CLINICAL TRIAL: NCT04943575
Title: Study to Evaluate the Efficacy of EZC Pak in Adults With Upper Respiratory Infection (URI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PPC Pharmaceuticals (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20214
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Active Comparator): EZC Pak
  Interventions: Dietary Supplement: EZC Pak
- Intervention 2 (Active Comparator): EZC Pak+D
  Interventions: Dietary Supplement: EZC Pak +D
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EZC Pak — After the onset of common cold symptoms, participants will take one pill (EZC Pak) each day for a period of 5 days.
  Arms: Intervention 1
Dietary Supplement: EZC Pak +D — After the onset of common cold symptoms, participants will take one pill (EZC Pak +D) each day for a period of 5 days.
  Arms: Intervention 2
Dietary Supplement: Placebo — After the onset of common cold symptoms, participants will take one pill (Placebo) each day for a period of 5 days.
  Arms: Placebo

SUMMARY:
A randomized-controlled interventional clinical trial to evaluate the effectiveness of EZC Pak & EZC Pak+D for the treatment of the common cold and/or a URI.

DETAILED DESCRIPTION:
This is a randomized-controlled interventional treatment study with three arms of comparable demographics to evaluate the efficacy of PPC Pharmaceuticals EZC Pak (& EZC Pak+D) to improve the severity and duration of the common cold or a URI in individuals. It is hypothesized that study participants will experience a positive impact on the duration and severity of their cold/URI while using EZC Pak (&EZC Pak+D). The second study objective is to examine if patients are accepting the test product as an alternative to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Seeking OTC remedies to reduce the severity and duration of their common cold symptoms, when they arise
* Must have a thermometer at home
* Must have a blood pressure monitor at home
* Ideally, uses one of the following devices: Apple Watch, Oura Ring, FitBit, other fitness trackers

Exclusion Criteria:

* Unwilling to try the test product for their cold
* Has any of the following medical conditions:

  * ragweed or daisy allergy
  * chronic seasonal allergies
  * liver disease
  * autoimmune or connective tissue disorder (e.g., rheumatoid arthritis, lupus, multiples sclerosis, HIV)
  * alcohol consumption more than 7 drinks per week, or more than 3 drinks per occasion
  * IV drug use
  * renal disease
  * females that are pregnant, want to become pregnant for the duration of the study, or who are breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Primary Objective: Reduction in severity of common cold symptoms | 6 months
  The primary objective of this study is to understand if EZC Pak (and EZC Pak +D) changes the severity and duration of an upper respiratory illness (URI) compared to a placebo. The study uses a scale of 1-4 (no symptoms to severe symptoms) to assess the effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, BSc, MSc, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radhakrishnan A, Spencer S, Yanamala N, Malepati S. Evaluating the Efficacy and Safety of EZC Pak, a 5-Day Combination Echinacea-Zinc-Vitamin C Dose Pack with or without Vitamin D, in the Management of Outpatient Upper Respiratory Infections. Infect Drug Resist. 2023 May 3;16:2561-2572. doi: 10.2147/IDR.S392087. eCollection 2023. PMID 37163146